CLINICAL TRIAL: NCT02080000
Title: Use of the R-wave to Optimise VV Delay in Heart Failure Patients Treated With Cardiac Resynchronisation Therapy
Brief Title: R-wave Optimisation in Cardiac Resynchronisation Therapy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROC001
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure, Systolic
Keywords: Heart Failure; Cardiac Resynchronisation Therapy; Biventricular Pacemaker; Optimisation
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimised V-V timing delay (Experimental): V-V timing delay setting on biventricular pacemaker will be optimised guided by size of R-wave on surface ECG
  Interventions: Other: Optimisation of V-V timing using R wave on surface ECG
- Standard V-V timing delay (Active Comparator): Standard settings
  Interventions: Other: Standard V-V timing settings

INTERVENTIONS:
Other: Optimisation of V-V timing using R wave on surface ECG
  Arms: Optimised V-V timing delay
Other: Standard V-V timing settings
  Arms: Standard V-V timing delay

SUMMARY:
The aim of this study is to investigate whether the use of a simple feature on the 12 lead electrocardiogram (ECG) to optimise pacemaker device programming can have clinically relevant benefit to patient management. More specifically it is to investigate whether using the R-wave in V1 of the surface ECG to guide the timings between left (LV) and right ventricular (RV) pacing improves response to Cardiac Resynchronisation Therapy.

ELIGIBILITY:
Inclusion Criteria

* The patient must have a biventricular pacemaker in situ, implanted for NYHA Class III / IV heart failure syndrome with impaired systolic function.
* Implantation indication must have included a left ventricular ejection fraction measured on transthoracic echo of <35% and either

  * a QRS duration of >150ms or
  * a QRS duration of 120 - 149ms with further evidence of dyssynchrony confirmed by echocardiography.
* Participants must have >95% true biventricular pacing over the 1 month before enrolment and throughout the observation period.
* The biventricular paced QRS complex morphology in lead V1 of subject's standard 12 lead surface ECG must show an R wave height of < 1mm or <20% of the total QRS deflection with standard LV offset settings applied.
* The subject's standard 12 lead surface ECG must show a right bundle branch block pattern in lead V1 during LV only pacing.
* The participant must be willing to comply with the protocol requirements including travelling to the Royal Bournemouth Hospital for the attendances required for the study and intend to have their long term device follow up at the Royal Bournemouth Hospital at the time of enrolment.
* Provision of informed consent Exclusion criteria
* Hypertrophic or restrictive cardiomyopathy
* Suspected acute myocarditis
* Correctable Valvulopathy
* An Acute Coronary Syndrome within the last 3 months
* Recent (within the last 3 months) or scheduled coronary revascularisation
* Treatment resistant hypertension
* Severe obstructive lung disease
* Pregnancy at the time of enrolment or a desire to become pregnant during the study period
* An inability to walk
* Reduced life expectancy not associated with cardiovascular disease (less than 1 year)
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Quality of Life Score | 3 months

SECONDARY OUTCOMES:
6 minute hall walk distance | 3 months
Left Ventricular End Systolic Volume Index | 3 months

OTHER OUTCOMES:
Hospitalisation for any cause | 3 months
Hospitalisation for Heart Failure | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom